CLINICAL TRIAL: NCT01161121
Title: Utilization of Lexiscan (Regadenoson)in the Cardiac Catheterization Lab to Achieve Maximal Hyperemia for Coronary Physiologic Assessment With Fractional Flow Reserve
Brief Title: Comparison of Intravenous Adenosine Infusion With Regadenoson Bolus for Inducing Maximal Coronary Hyperemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: University of Florida (Other); Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Michael J. Lim, Director, Division of Cardiology, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rega-9I06
Record Dates: First submitted 2010-07-06; First posted 2010-07-13 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: Fractional flow reserve; adenosine; regadenoson
MeSH Terms: conditions — Coronary Artery Disease | interventions — Adenosine; regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adenosine then Regadenoson (Experimental): Adenosine infusion will be compared to Regadenoson for efficacy and safety/side effects. Arterial blood pressure, coronary pressure, heart rate, oxygen saturation and coronary flow, FFR, and coronary flow velocity will be assessed. Safety will be assessed by monitoring for any side effects such as chest pain, headache, flushing, nausea, or arrhythmias. Adenosine infusion will be administered at 140 mcg/kg for 2 minutes and once mean coronary flow velocity returns to within 15% of pre-dose value, Regadenoson IV bolus 0.4 mg/5 ml will be administered followed by a 5 cc normal saline flush.
  Interventions: Drug: adenosine; Drug: regadenoson

INTERVENTIONS:
Drug: adenosine — Measuring FFR and Coronary Flow Reserve after administration of IV adenosine 140 mcg/kg/min for 2 minutes.
  Other Names: Adenoscan(adenosine)
Drug: regadenoson — Measuring FFR and Coronary Flow Reserve after administration of IV regadenoson 0.4 mg over 10 seconds.
  Other Names: Lexiscan

SUMMARY:
The purpose of this study is to determine if regadenoson is as safe and effective as adenosine when used in the cardiac catheterization lab during measurement of coronary flow reserve and fractional flow reserve. The study hypothesis is the assessment of Fractional Flow Reserve (FFR) in the catheterization lab can be performed with equivalent accuracy when hyperemia is induced with IV Regadenoson compared with IV Adenosine without compromising patient safety.

DETAILED DESCRIPTION:
Patients with clinical indications to be assessed by fractional flow reserve (FFR) will be included. Following diagnostic angiography in the catheterization lab, the patient will have a guide catheter placed in the artery to be assessed followed by placing a pressure guidewire down the coronary vessel and past the lesion of interest. FFR will be measured in the traditional manner, with intravenous adenosine infusing at 140 mcg/kg/min until maximal steady state hyperemia is reached. At this point, the FFR will be recorded as Pd (distal pressure from the pressure wire in the coronary artery) divided by Pa (proximal pressure from the guide catheter). The adenosine infusion will then be stopped and the patient's hemodynamics allowed to return to baseline. Once baseline state is again achieved, an intravenous bolus of regadenson (0.4 mg) will be given and FFR will be remeasured as the lowest steady state Pd/Pa. Patients will be enrolled at two sites, The University of Florida - where FFR will be measured alone, and Saint Louis University, where coronary flow will be measured simultaneously to evaluate the effect of regadenoson on coronary flow velocity as compared to adenosine. The primary endpoint of the study will be to compare the FFR achieved with adeonsine to that obtained with regadenoson.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients greater than 18 years old (If female, pt. must be post-menopausal, surgically sterile, or be non-pregnant as determined by a negative urine or serum beta human chorionic gonadotropin (B-HCG) pregnancy test within 24 hours prior to enrollment.
* Provided written consent approved by Institutional Review Board and provided Health Insurance Portability and Accountability Act (HIPAA) authorization
* Have at least one coronary stenosis (greater or equal to 40% but less than 70& narrowing by visual inspection) and technically accessible coronary artery into which the pressure wire may be introduced.

Exclusion Criteria:

* ST elevation myocardial infarction
* Cardiogenic shock
* Pregnancy
* Total vessel occlusion
* Extremely tortuous coronary arteries
* Second and third degree heart block without pacemaker
* Severe chronic obstructive pulmonary disease and active bronchospasm
* Less than age 18 years
* Have received theophylline, aminophylline, pentoxifylline or dipyridamole within 12 hours of FFR measurement.
* Has severe 3 vessel disease defined by >80% luminal narrowing by visual inspection
* Known hypersensitivity to adenosine or regadenoson
* Recent uncontrolled ventricular arrhythmia
* History of greater than Type I atrioventricular block, symptomatic resting bradycardia, sick sinus syndrome (without permanent pacemaker)
* History of heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Lim, MD, Principal Investigator — St. Louis University
Locations (2):
- United States (2):
  - University of Florida, Jacksonville, Florida
  - St. Louis University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pijls NH, Van Gelder B, Van der Voort P, Peels K, Bracke FA, Bonnier HJ, el Gamal MI. Fractional flow reserve. A useful index to evaluate the influence of an epicardial coronary stenosis on myocardial blood flow. Circulation. 1995 Dec 1;92(11):3183-93. doi: 10.1161/01.cir.92.11.3183. PMID 7586302
- [Background] Iskandrian AE, Bateman TM, Belardinelli L, Blackburn B, Cerqueira MD, Hendel RC, Lieu H, Mahmarian JJ, Olmsted A, Underwood SR, Vitola J, Wang W; ADVANCE MPI Investigators. Adenosine versus regadenoson comparative evaluation in myocardial perfusion imaging: results of the ADVANCE phase 3 multicenter international trial. J Nucl Cardiol. 2007 Sep-Oct;14(5):645-58. doi: 10.1016/j.nuclcard.2007.06.114. PMID 17826318
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Lim MJ, Kern MJ. Coronary pathophysiology in the cardiac catheterization laboratory. Curr Probl Cardiol. 2006 Aug;31(8):493-550. doi: 10.1016/j.cpcardiol.2006.04.002. PMID 16920478
- [Derived] Stolker JM, Lim MJ, Shavelle DM, Morris DL, Angiolillo DJ, Guzman LA, Kennedy KF, Weber E, Zareh M, Neumayr RH, Zenni MM. Pooled comparison of regadenoson versus adenosine for measuring fractional flow reserve and coronary flow in the catheterization laboratory. Cardiovasc Revasc Med. 2015 Jul-Aug;16(5):266-71. doi: 10.1016/j.carrev.2015.05.011. Epub 2015 Jun 5. PMID 26242981

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients provided written consent for participation in the study prior to cardiac catheterization. Diagnostic coronary angiography was performed utilizing standard techniques. Patients in whom the operator believed needed physiologic coronary assessment with Fractional Flow Reserve (FFR) were then eligible for participation in the study.
Groups:
- Adenosine Then Regadenoson: Adenosine infusion will be compared to Regadenoson for efficacy and safety/side effects. Arterial blood pressure, coronary pressure, heart rate, oxygen saturation and coronary flow, FFR, and coronary flow velocity will be assessed. Safety will be assessed by monitoring for any side effects such as chest pain, headache, flushing, nausea, or arrhythmias. All patients to receive Adenosine infusion followed by Regadenoson IV bolus upon return of coronary flow velocity to 15% of pre-dose value.
  Adenosine : Injection of IV Adenosine for 2 minutes at rate of 140mcg/kg to dilate coronary arteries and provoke maximal hyperemia.
  Regadenoson : Administration of IV regadenoson bolus 0.4 mg/5 mls over 10 seconds followed by a 5 cc NS saline flush
Period: Overall Study
Arm/Group | Adenosine Then Regadenoson
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with intermediate to severe, single vessel or multi-vessel, angiographic coronary artery disease(visual 40%-70% angiographic stenosis) whose lesion assessment with FFR is planned, were eligible for enrollment. A total of up to 50 subjects(25 at University of Florida Health Science Center and 25 at St. Louis University) will be enrolled.
Groups:
- Adenosine, Regadenoson: Each patient underwent standard intravenous adenosine infusion (140mcg/kg/min) with invasive pressure recordings for 2 min, or until maximal hyperemia occurred. Five minutes after return to baseline hemodynamics, a single intravenous bolus of 0.4 mg regadenoson was administered, and pressures were recorded for 5 min. FFR values were compared by linear regression and Bland-Altman analysis.
Arm/Group | Adenosine, Regadenoson
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Difference in FFR Between IV Adenosine and IV Regadenoson
Description: FFR (as calculated by the ratio of lowest Pd/Pa at maximal hyperemia) was compared between hyperemia achieved with adenosine and with regadenoson
Time Frame: At maximal, steady-state hyperemia
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ratio (Pd/Pa)
Groups:
- Adenosine: Adenosine infusion will be compared to Regadenoson for safety/side effects. Arterial blood pressure, coronary pressure, heart rate, oxygen saturation and coronary flow, FFR, and coronary flow velocity will be assessed. Safety will be assessed by monitoring for any side effects such as chest pain, headache, flushing, nausea, or arrhythmias.
  Adenosine : Injection of IV Adenosine for 2 minutes at rate of 140mcg/kg to dilate coronary arteries and provoke maximal hyperemia
- Regadenoson: Once the mean coronary flow velocity returns to within 15% pre-dose value following IV infusion of Adenosine, Regadenoson IV injection will be given at 0.4 mg 5/ml- 0.08mg/ml over 10 seconds followed by a 5 cc IV saline flush.
  regadenoson : Measuring FFR and Coronary Flow Reserve after administration of IV regadenoson 0.4 mg over 10 seconds.
Arm/Group | Adenosine | Regadenoson
Number analyzed (Participants) | 46 | 46
ratio (Pd/Pa) | 0.84 (0.11) | 0.84 (0.10)

2. Secondary Outcome: Heart Rate Changes With Drug
Description: Maximal heart rate documented following the administration of each agent
Time Frame: During drug infusion and until restoration of baseline hemodynamics
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Adenosine: With infusion of 140 mcg/kg/min
- Regadenosine: With bolus infusion of 0.4 mg
Arm/Group | Adenosine | Regadenosine
Number analyzed (Participants) | 46 | 46
beats per minute
  Baseline Heart Rate | 70.8 (11.5) | 72.4 (12.0)
  Maximal Heart Rate | 81.7 (13.4) | 90.4 (13.0)

3. Secondary Outcome: Side Effects of Medication Administration
Description: Chest pain, chest discomfort, burning, flushing, headache, nausea, or shortness of breath
Time Frame: During drug infusion and until restoration of baseline hemodynamics
Measure: Number; unit: participants
Arm/Group | Adenosine | Regadenoson
Number analyzed (Participants) | 46 | 46
participants
  Dyspnea | 14 | 13
  Chest Pain | 16 | 13
  Any Symptom | 27 | 28

ADVERSE EVENTS:
Groups:
- Adenosine: Adenosine infusion will be compared to Regadenoson for safety/side effects. Arterial blood pressure, coronary pressure, heart rate, oxygen saturation and coronary flow, FFR, and coronary flow velocity will be assessed. Safety will be assessed by monitoring for any side effects such as chest pain, headache, flushing, nausea, or arrhythmias.
  Adenosine : Injection of IV Adenosine for 2 minutes at rate of 140mcg/kg to dilate coronary arteries and provoke maximal hyperemia
  adenosine : Measuring FFR and Coronary Flow Reserve after administration of IV adenosine 140 mcg/kg/min for 2 minutes.
  regadenoson : Measuring FFR and Coronary Flow Reserve after administration of IV regadenoson 0.4 mg over 10 seconds.
- Regadenoson: Once the mean coronary flow velocity returns to within 15% pre-dose value then Regadenoson IV injection will be given at 0.4 mg 5/ml- 0.08mg/ml. Then, a 5 cc saline flush will be administered.
  regadenoson : Measuring FFR and Coronary Flow Reserve after administration of IV regadenoson 0.4 mg over 10 seconds.
Arm/Group | Adenosine | Regadenoson
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 27/46 | 28/46
OTHER ADVERSE EVENTS (reported when occurring in more than 2.17% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adenosine (N=46) | Regadenoson (N=46)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 13 (13)
Flushing (Skin and subcutaneous tissue disorders) | 6 (6) | 9 (9)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Cardiac General -Chest Pain (Cardiac disorders) | 16 (16) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less